CLINICAL TRIAL: NCT00007202
Title: A Pilot Open-Label Phase II Clinical Trial to Evaluate the Safety and Efficacy of a Compact Three Drug Antiretroviral Treatment Regimen for Subjects With Acute HIV-1 Infection or Recent HIV-1 Seroconversion
Brief Title: Safety and Effectiveness of a Three-Drug Combination Treatment for Recently Infected or Converted HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: AI-03-005; 10431 (Registry Identifier: DAIDS ES); AIEDRP AI-03-005; Substudy AI-03-006; Substudy AI-03-007; Substudy AI-03-008
Record Dates: First submitted 2000-12-15; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Virus Replication; HIV-1; Didanosine; Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Sensitivity and Specificity; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Reverse Transcriptase Polymerase Chain Reaction; Acute Infection
MeSH Terms: conditions — HIV Infections; Hypersensitivity | interventions — Atazanavir Sulfate; Stavudine; Didanosine

INTERVENTIONS:
Drug: Atazanavir
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of stavudine (d4T), didanosine (ddI), and BMS-232632 when given early in the course of HIV infection.

Acute HIV infection may develop in patients that are exposed to the HIV virus. Following infection, the viral load (level of HIV in the blood) rises rapidly over the next few days to weeks. It is not known which is the best treatment in patients with very early HIV infection. Researchers believe these patients may respond well to strong early treatment. A combination consisting of enteric-coated didanosine (ddI-EC), stavudine (d4T), and the HIV-1 protease inhibitor, BMS-232632, will be tested.

DETAILED DESCRIPTION:
Acute primary HIV-1 infection (PHI) follows exposure to the HIV-1 virus and results in a rapid rise in plasma viremia within days to 1 to 3 weeks. Individuals with acute PHI or early HIV-1 infection represent a potentially unique patient population in which to evaluate potent antiretroviral therapies because of the degree of viral heterogeneity and the fact that immunologic disruption is likely to be lower than in later stages of HIV-1 disease. The optimal treatment for acute PHI is unknown. This study evaluates a regimen consisting of enteric-coated didanosine (ddI-EC), stavudine (d4T), and the HIV-1 protease inhibitor, BMS-232632.

Patients are enrolled into Group I or Group II and may participate in substudies. Patients in Group I receive ddI-EC, d4T, and BMS-232632 daily for 52 weeks. Clinical, virologic, and immunologic evaluations are performed on Days 2, 7, 14, 21, and 28, then every 4 weeks through Week 24, and then every 8 weeks thereafter through Week 48. Based on laboratory results from the Week 48 visit, a decision is made by Week 52 whether or not to continue study medications for an additional 52 weeks. Evaluation schedules for those patients enrolled in substudies may be different. Group II patients elect not to receive antiretroviral treatment and are followed as a natural history disease group to be compared with patients in Group I. They are followed according to the same schedule of evaluations as those enrolled in Group I, unless otherwise specified as part of their participation in substudies. All patients are followed in this study at 8-week intervals for a total duration of 104 weeks (2 years). HIV will be measured in plasma and tissues to determine reduction in replication for a duration of at least 48 weeks.

The 3 substudies in which patients may participate are AI-03-006, Lymphoid Tissue Substudy; AI-03-007, Immunology Substudy of cytolytic and co-stimulatory markers, T-cell repertoire, and cytokine and chemokine elaboration; and AI-03-008, Viral Dynamics and Diversity Substudy.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have early HIV infection or show recent seroconversion (going from HIV-negative to HIV-positive).
* Are at least 18 years old.
* Agree to 2 barrier methods of birth control, if heterosexually active men or women, during the study and for 3 months after.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have received prior antiretroviral therapy.
* Have received interferons, interleukins, colony-stimulating factors, radiation, cytotoxic chemotherapy, or HIV vaccines within 30 days prior to study entry.
* Have had any experimental therapy within 30 days prior to study entry.
* Are pregnant or breast-feeding.
* Patients will not be eligible for Group I if they:
* Have had pancreatitis (inflammation of the pancreas).
* Have received alpha tocopherol (vitamin E), amiodarone, astemizole, carbamazepine, cisapride, ergotamine/diergotamine, estrogens, fluvastatin, glucocorticoids, itraconazole, ketoconazole, midazolam, phenobarbital, phenytoin, quinidine, rifampin, rifabutin, sildenafil, statin drugs (simvastatin, pravastatin, atorvastatin) used for reduction of triglyceride or cholesterol levels, terfenadine, triazolam, or warfarin within 14 days of study entry.
* Have received chloramphenicol, cisplatin, clioquinol, dapsone, diphenylhydantoin, disulfiram, ethionamide, glutethimide, gold, hydralazine, isoniazid, metronidazole, pyridoxine, sodium cyanate, thalidomide, vincristine, or zalcitabine within 30 days of study entry. In certain cases, patients taking these drugs may still be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constance Benson, Study Chair; Robert Schooley, Study Chair; Wheaton Williams, Study Chair
Locations (5):
- United States (4):
  - Univ. of Colorado Health Sciences Ctr. AIEDRP, Denver, Colorado
  - AIDS Research Consortium of Atlanta, Inc. (ARCA) AIEDRP CRS, Atlanta, Georgia
  - Feinberg School of Medicine, HIV/ACTU AIEDRP CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr., Dept. of Infectious Disease AIEDRP CRS, Chicago, Illinois
- Centro de Referencia Estadual de AIDS AIEDRP, Salvador, Estado de Bahia, Brazil